CLINICAL TRIAL: NCT01550198
Title: Early Detection of Shock in Critically Ill Newborn Infants. The Impact of Advanced Hemodynamic Monitoring
Brief Title: Early Detection of Neonatal Shock
Acronym: Edscini
Status: Terminated | Type: Observational
Why Stopped: Problems with availability of cardiac output monitoring system
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Edscini Study 1.0
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Impact of Advanced Hemodynamic Monitoring
Keywords: newborn; shock; hemodynamics; cardiac output; blood pressure
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Newborns: Critically ill newborns admitted to level III neonatal intensive care unit of a university hospital, who will be monitored using transpulmonary ultrasound dilution ("advanced hemodynamic monitoring")
  Interventions: Device: Advanced hemodynamic monitoring

INTERVENTIONS:
Device: Advanced hemodynamic monitoring — Comprehensive advanced hemodynamic monitoring

SUMMARY:
The purpose of this study is to evaluate the hypothesis that advanced hemodynamic monitoring results in an earlier detection of circulatory failure in newborn infants

ELIGIBILITY:
Inclusion Criteria:

* Birth weight >700 grams
* Arterial catheter in place
* Central venous catheter in place
* Informed consent from parents/legal representatives

Exclusion Criteria:

* Life-threatening congenital defects
* Congenital heart defects, except patent ductus arteriosus and patent foramen ovale

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neonates admitted to a neonatal intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2021-12 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Cardiac output assessed by transpulmonary ultrasound dilution and simultaneously clinically estimated cardiac output | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Willem de Boode, MD PhD, Principal Investigator — Radboud University Nijmegen Medical Center, Nijmegen, The Netherlands
Locations (1):
- Radboud University Nijmegen Medical Centre, Department of Neonatology, Nijmegen, Netherlands